CLINICAL TRIAL: NCT01837862
Title: A Phase I Study of Mebendazole for the Treatment of Pediatric Gliomas
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Julie Krystal (Other)
Collaborators: Janssen Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Julie Krystal, Head, Developmental Therapeutics, Northwell Health
Organization: Northwell Health (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCMC1411
Record Dates: First submitted 2013-04-16; First posted 2013-04-23 (Estimated); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Pilomyxoid Astrocytoma; Pilocytic Astrocytoma; Glioma, Astrocytic; Optic Nerve Glioma; Pleomorphic Xanthoastrocytoma; Glioblastoma Multiforme; Anaplastic Astrocytoma; Gliosarcoma; Diffuse Intrinsic Pontine Glioma; DIPG; Low-grade Glioma; Brainstem Glioma
Keywords: pilomyxoid astrocytoma; Pilocytic Astrocytoma; Glioma; Optic Nerve Glioma; mebendazole; Pleomorphic Xanthoastrocytoma; glioblastoma multiforme; anaplastic astrocytoma; gliosarcoma; diffuse intrinsic pontine glioma; DIPG; low-grade glioma; high-grade glioma; brainstem glioma; pediatric
MeSH Terms: conditions — Astrocytoma; Optic Nerve Glioma; Glioblastoma; Gliosarcoma; Diffuse Intrinsic Pontine Glioma; Glioma | interventions — Mebendazole; Vincristine; Carboplatin; Temozolomide; Bevacizumab; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low-grade Glioma (Experimental): Patients on the low-grade arm will receive treatment with seven 10-week cycles of carboplatin, vincristine, temozolomide, and mebendazole.
  Interventions: Drug: Mebendazole; Drug: Vincristine; Drug: Carboplatin; Drug: Temozolomide
- High-grade Glioma/Pontine Glioma (Experimental): Patients on the high-grade glioma/pontine glioma arm will receive treatment with twelve 28-day cycles of bevacizumab, irinotecan, and mebendazole.
  *High grade arm enrollment complete, no additional spots
  Interventions: Drug: Mebendazole; Drug: Bevacizumab; Drug: Irinotecan

INTERVENTIONS:
Drug: Mebendazole — Mebendazole will be given orally twice daily for over the course of treatment (70 weeks for low-grade glioma patients, 48 weeks for high-grade glioma/pontine glioma patients). Mebendazole will be prescribed according to the particular dose cohort for each patient (50 mg/kg/day, 100 mg/kg/day, or 200 mg/kg/day).
  Other Names: Vermox
Drug: Vincristine — Low-grade glioma patients only. Vincristine will be dosed as per the following: For patients < 12kg: 0.05 mg/kg; for patient > 12kg: 1.5mg/m2 (maximal dose 2.0 mg). Vincristine will be administered intravenously on Day 1 of weeks 0,1,2,3,4,5 during the 10-week induction cycle and on Day 1 of Weeks 0,1,2 of the six 10-week maintenance cycles.
  Other Names: Oncovin
  Arms: Low-grade Glioma
Drug: Carboplatin — Low-grade glioma patients only. Carboplatin will be dosed at 175 mg/m2. Carboplatin will be administered intravenously on Day 1 of Weeks 0,1,2,3 of the 10-week Induction cycle, and on Day 1 of Weeks 0,1,2,3 during the six 10-week maintenance cycles.
  Other Names: Paraplatin
  Arms: Low-grade Glioma
Drug: Temozolomide — Low-grade glioma patients only. Temozolomide will be dosed at 200 mg/m2/day. Temozolomide will be given orally for 5 days during Week 6 of the 10-week induction cycle and for 5 days during Week 6 of the six 10-week maintenance cycles.
  Other Names: Temodar
  Arms: Low-grade Glioma
Drug: Bevacizumab — High-grade glioma/pontine glioma patients only. Bevacizumab will be dosed at 10mg/kg/dose. Bevacizumab will be administered intravenously on Days 1 and 15 of each maintenance cycle.
  Other Names: Avastin
  Arms: High-grade Glioma/Pontine Glioma
Drug: Irinotecan — High-grade glioma/pontine glioma patients only. Irinotecan will be administered at doses 125 mg/m2, 150 mg/m2, 250 mg/m2, or 300 mg/m2, depending on patient tolerance and concomitant enzyme-inducing anti-epileptic medication use. Irinotecan will be administered intravenously on Days 1 and 15 of each maintenance cycle.
  Other Names: CPT-11; Camptosar
  Arms: High-grade Glioma/Pontine Glioma

SUMMARY:
This is a study to determine the safety and efficacy of the drug, mebendazole, when used in combination with standard chemotherapy drugs for the treatment of pediatric brain tumors. Mebendazole is a drug used to treat infections with intestinal parasites and has a long track record of safety in humans. Recently, it was discovered that mebendazole may be effective in treating cancer as well, in particular brain tumors. Studies using both cell cultures and mouse models demonstrated that mebendazole was effective in decreasing the growth of brain tumor cells.

This study focuses on the treatment of a category of brain tumors called gliomas. Low-grade gliomas are tumors arising from the glial cells of the central nervous system and are characterized by slower, less aggressive growth than that of high-grade gliomas. Some low-grade gliomas have a more aggressive biology and an increased likelihood of resistance or recurrence.

Low-grade gliomas are often able to be treated by observation alone if they receive a total surgical resection. However, tumors which are only partially resected and continue to grow or cause symptoms, or those which recur following total resection require additional treatment, such as chemotherapy. Due to their more aggressive nature, pilomyxoid astrocytomas, even when totally resected, will often be treated with chemotherapy. The current first-line treatment at our institution for these low-grade gliomas involves a three-drug chemotherapy regimen of vincristine, carboplatin, and temozolomide. However, based on our data from our own historical controls, over 50% of patients with pilomyxoid astrocytomas will continue to have disease progression while on this treatment. We believe that mebendazole in combination with vincristine, carboplatin, and temozolomide may provide an additional therapeutic benefit with increased progression-free and overall survival for low-grade glioma patients, particularly for those with pilomyxoid astrocytomas.

High grade gliomas are more aggressive tumors with poor prognoses. The standard therapy is radiation therapy. A variety of adjuvant chemotherapeutic combinations have been used, but with disappointing results. For high-grade gliomas this study will add mebendazole to the established combination of bevacizumab and irinotecan to determine this combinations safety and efficacy

DETAILED DESCRIPTION:
This is a phase I/II study of mebendazole in combination with standard of care agents for pediatric patients with gliomas. Patients with low-grade gliomas will receive a regimen of mebendazole in combination with vincristine, carboplatin, and temozolomide. Patients with high-grade gliomas and diffuse intrinsic pontine gliomas will receive a regimen of mebendazole in combination with bevacizumab and irinotecan. Surgical resection of the tumor will be attempted initially with the goal of achieving a gross total resection without substantial neurologic deficit. Subtotal resection may be preferable depending on the location of the tumor. Optic pathway gliomas and diffuse intrinsic pontine gliomas may remain unresected. Patients with high-grade gliomas or diffuse intrinsic pontine gliomas will undergo local irradiation of their tumor before beginning protocol treatment. Low-grade glioma patients will not receive radiation therapy. Patients who have been previously treated with chemotherapy will be eligible for the study provided they have not previously failed therapy with any of the chemotherapeutic agents.

Patients with eligible tumors will be consented for enrollment into the study. The study patients will be divided into two groups (low-grade glioma and high-grade/pontine glioma) for the purpose of determining the maximally tolerated dose of mebendazole. These two groups will be treated independently with regard to patient accrual, dose escalation, and evaluation of toxicity. In addition to their standard chemotherapy regimen, patients in both cohorts will receive mebendazole. Mebendazole doses will be escalated from the initial dose level of 50 mg/kg/day divided twice daily, to a second dose level of 100 mg/kg/day divided twice daily, to the final dose level of 200 mg/kg/day divided twice daily, in cohorts of three patients per dose level. A standard "3+3" design will be used for determining dose escalation.

Phase I safety monitoring for the low-grade group will take place during a trial period beginning with start of therapy and ending following the tenth week of induction therapy. Phase I safety monitoring for the high-grade/pontine glioma group will take place during a trial period beginning with the start of maintenance therapy through the twelfth week of maintenance therapy (3 cycles).

After determination of maximally tolerated dose for each group, the study will continue to evaluate efficacy of this regimen. The study will be amended for the maximally tolerated dose for each group to be used in the remainder of the study. Patients currently on study will continue with maintenance therapy. To document the degree of residual tumor, standard whole brain MRI with and without contrast (gadolinium) will be performed following a specified intervals. Following completion of therapy, patients will continue to be monitored by MRI to assess progression-free and overall-survival.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 1 year of age and ≤ 21 years of age
2. Diagnosis

   2.1. Group A - Low-grade Glioma Group:

   Histology: Biopsy-proven:
   * Pilocytic Astrocytoma
   * Fibrillary Astrocytoma
   * Pilomyxoid Astrocytoma
   * Pleomorphic Xanthoastrocytoma
   * Other low grade astrocytomas

   Children with optic pathway tumors must have evidence of progressive disease on MRI and/or symptoms of deteriorating vision or, progressive hypothalamic/pituitary dysfunction or, diencephalic syndrome or precocious puberty.

   Patients with relapsed low-grade gliomas who have been previously treated with chemotherapy will be eligible for the study provided they have not previously failed therapy with any of the chemotherapeutic agents used in this study.

   2.2 Group B - High-grade Glioma/Pontine Glioma Group:

   Histology: Biopsy-proven
   * Anaplastic astrocytoma
   * Glioblastoma multiforme
   * Gliosarcoma.

   Patients with primary spinal cord malignant gliomas are eligible.

   For primary brainstem tumors, histologic verification is not required. Patients are eligible when diagnosed with clinical and radiographic (MRI) evidence of tumors which diffusely involve the brainstem. Patients with tumors which intrinsically (greater than 50% intra-axial) involve the pons or pons and medulla or pons and midbrain or entire brainstem are eligible. Tumors may contiguously involve the thalamus or upper cervical cord.
3. Timing of therapy:

   Patients must be enrolled before treatment begins. Treatment must start within 14 days of study enrollment.

   All clinical and laboratory studies to determine eligibility must be performed within 7 days prior to enrollment unless otherwise indicated in the eligibility section.
4. Adequate hematologic, renal, liver function as demonstrated by laboratory values.
5. Negative pregnancy test in women of childbearing potential within 7 days of initiating investigational therapy
6. Life expectancy ≥ 3 months
7. Concurrent medications: It is recommended that patients are weaned off or are on a tapering dose of corticosteroids before starting therapy on study.
8. Patient or legal guardian must give written, informed consent or assent (when applicable)
9. Recent mothers must agree not to breast feed while receiving medications on study.

Exclusion criteria:

1. Age < 1 year or > 21 years
2. Patients who have known allergy to mebendazole or benzimidazole class drugs.
3. Patients who have previously had a severe side effect, such as agranulocytosis and neutropenia, in conjunction with previous mebendazole or benzimidazole class drug for a parasitic infection .
4. Patients who are taking metronidazole and cannot be safely moved to a different antibiotic greater than 7 days prior to starting mebendazole therapy.
5. Pregnant female patients are not eligible for this study. Pregnancy tests with a negative result must be obtained in all post-menarchal females.
6. Lactating females must agree they will not breastfeed a child while on this study.
7. Males and females of reproductive potential may not participate unless they agree to use an effective contraceptive method and continue to do so for at least 6 months after the completion of therapy.
8. Patients who are unable to take oral medications because of significant vomiting will be excluded.
9. Group A - Low-grade Glioma Group ONLY:

   Patients who have failed prior chemotherapy with vincristine, carboplatin, or temozolomide for this tumor are excluded.

   Patients with Neurofibromatosis Type 1
10. Group B - High-grade Glioma/Pontine Glioma Group ONLY:

Patients who failed prior chemotherapy with bevacizumab or irinotecan for this tumor are excluded.

Patients who progressed on or within 12 weeks after completion of radiotherapy are excluded.

Patients with a history or current condition that would preclude the use of bevacizumab

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Estimated)
Dates: Start 2013-10-22 (Actual); Primary Completion 2024-04 (Actual); Study Completion 2024-04 (Actual)

PRIMARY OUTCOMES:
Maximally tolerated dose of mebendazole in combination with vincristine, carboplatin, and temozolomide | Assessed after the 10 week Induction cycle
  Low-grade glioma patients will receive an assigned dose of mebendazole twice daily in combination with vincristine, carboplatin and temozolomide. During a 10 week induction period, patients will be assessed for dose-limiting toxicity that is beyond the expected toxicity from the standard regimen of vincristine, carboplatin, and temozolomide alone. This outcome measure will use a standard 3+3 design to dose-escalate mebendazole in three dose cohorts of 50 mg/kg/day, 100 mg/kg/day, and 200 mg/kg/day.
Maximally tolerated dose of mebendazole in combination with bevacizumab and irinotecan. | Assessed after the first 3 maintenance cycles (12 weeks)
  High-grade glioma/pontine glioma patients will receive an assigned dose of mebendazole twice daily in combination with bevacizumab and irinotecan. During the first three maintenance therapy cycles (12 weeks), patients will be assessed for dose-limiting toxicity that is beyond the expected toxicity from the standard regimen of bevacizumab and irinotecan alone. This outcome measure will use a standard 3+3 design to dose-escalate mebendazole in three dose cohorts of 50 mg/kg/day, 100 mg/kg/day, and 200 mg/kg/day.

SECONDARY OUTCOMES:
Survival of patients with low-grade gliomas | 3-years post-treatment
  3-year event-free survival (EFS) and overall survival (OS) of patients with low-grade gliomas treated with carboplatin, vincristine, temozolomide, and mebendazole in combination following surgical resection, to the extent feasible.
Survival of patients with high-grade gliomas | 3-years post-treatment
  3-year event-free survival (EFS) and overall survival (OS) of patients with high-grade gliomas treated with bevacizumab, irinotecan, and mebendazole in combination following surgical resection to the extent feasible and local irradiation.
Frequency of cerebrospinal fluid (CSF) dissemination in pilomyxoid astrocytoma | 3 years post-treatment
  The frequency of tumor dissemination in the CSF of patients with pilomyxoid astrocytomas treated with carboplatin, vincristine, temozolomide, and mebendazole.
Partial or complete response rate on MRI of patients with high-grade gliomas/pontine gliomas | 3-years post-treatment
  The percentage of patients demonstrating a partial (greater than 50% decrease in tumor volume in 3 dimensions) or complete response on MRI in patients with high-grade gliomas treated with mebendazole in combination with bevacizumab and irinotecan, after surgical resection, to the extent feasible and local irradiation.
Partial or complete response rate on MRI of patients with low-grade gliomas | 3-years post-treatment
  The percentage of patients demonstrating a partial (greater than 50% decrease in tumor volume in 3 dimensions) or complete response on MRI in patients with low-grade gliomas treated with mebendazole in combination with vincristine, carboplatin and temozolomide after surgical resection, to the extent feasible.

CONTACTS AND LOCATIONS:
Overall Officials: Julie Krystal, MD, Principal Investigator — Northwell Health
Locations (1):
- Cohen Children's Medical Center of New York, New Hyde Park, New York, United States

REFERENCES:
- [Background] Tihan T, Fisher PG, Kepner JL, Godfraind C, McComb RD, Goldthwaite PT, Burger PC. Pediatric astrocytomas with monomorphous pilomyxoid features and a less favorable outcome. J Neuropathol Exp Neurol. 1999 Oct;58(10):1061-8. doi: 10.1097/00005072-199910000-00004. PMID 10515229
- [Background] Komotar RJ, Mocco J, Jones JE, Zacharia BE, Tihan T, Feldstein NA, Anderson RC. Pilomyxoid astrocytoma: diagnosis, prognosis, and management. Neurosurg Focus. 2005 Jun 15;18(6A):E7. PMID 16048293
- [Background] Paraskevopoulos D, Patsalas I, Karkavelas G, Foroglou N, Magras I, Selviaridis P. Pilomyxoid astrocytoma of the cervical spinal cord in a child with rapid progression into glioblastoma: case report and literature review. Childs Nerv Syst. 2011 Feb;27(2):313-21. doi: 10.1007/s00381-010-1171-5. Epub 2010 May 12. PMID 20461521
- [Background] Komotar RJ, Carson BS, Rao C, Chaffee S, Goldthwaite PT, Tihan T. Pilomyxoid astrocytoma of the spinal cord: report of three cases. Neurosurgery. 2005;56(1):191. doi: 10.1227/01.NEU.0000146212.95421.B3. PMID 15617606
- [Background] Bauman G, Lote K, Larson D, Stalpers L, Leighton C, Fisher B, Wara W, MacDonald D, Stitt L, Cairncross JG. Pretreatment factors predict overall survival for patients with low-grade glioma: a recursive partitioning analysis. Int J Radiat Oncol Biol Phys. 1999 Nov 1;45(4):923-9. doi: 10.1016/s0360-3016(99)00284-9. PMID 10571199
- [Background] Desai KI, Nadkarni TD, Muzumdar DP, Goel A. Prognostic factors for cerebellar astrocytomas in children: a study of 102 cases. Pediatr Neurosurg. 2001 Dec;35(6):311-7. doi: 10.1159/000050443. PMID 11786699
- [Background] Gajjar A, Sanford RA, Heideman R, Jenkins JJ, Walter A, Li Y, Langston JW, Muhlbauer M, Boyett JM, Kun LE. Low-grade astrocytoma: a decade of experience at St. Jude Children's Research Hospital. J Clin Oncol. 1997 Aug;15(8):2792-9. doi: 10.1200/JCO.1997.15.8.2792. PMID 9256121
- [Background] Wisoff JH, Boyett JM, Berger MS, Brant C, Li H, Yates AJ, McGuire-Cullen P, Turski PA, Sutton LN, Allen JC, Packer RJ, Finlay JL. Current neurosurgical management and the impact of the extent of resection in the treatment of malignant gliomas of childhood: a report of the Children's Cancer Group trial no. CCG-945. J Neurosurg. 1998 Jul;89(1):52-9. doi: 10.3171/jns.1998.89.1.0052. PMID 9647172
- [Background] Finlay JL, Wisoff JH. The impact of extent of resection in the management of malignant gliomas of childhood. Childs Nerv Syst. 1999 Nov;15(11-12):786-8. doi: 10.1007/s003810050471. PMID 10603023
- [Background] Pollack IF, Claassen D, al-Shboul Q, Janosky JE, Deutsch M. Low-grade gliomas of the cerebral hemispheres in children: an analysis of 71 cases. J Neurosurg. 1995 Apr;82(4):536-47. doi: 10.3171/jns.1995.82.4.0536. PMID 7897512
- [Background] Packer RJ, Ater J, Allen J, Phillips P, Geyer R, Nicholson HS, Jakacki R, Kurczynski E, Needle M, Finlay J, Reaman G, Boyett JM. Carboplatin and vincristine chemotherapy for children with newly diagnosed progressive low-grade gliomas. J Neurosurg. 1997 May;86(5):747-54. doi: 10.3171/jns.1997.86.5.0747. PMID 9126887
- [Background] Conway PD, Oechler HW, Kun LE, Murray KJ. Importance of histologic condition and treatment of pediatric cerebellar astrocytoma. Cancer. 1991 Jun 1;67(11):2772-5. doi: 10.1002/1097-0142(19910601)67:113.0.co;2-#. PMID 1851047
- [Background] Fisher BJ, Leighton CC, Vujovic O, Macdonald DR, Stitt L. Results of a policy of surveillance alone after surgical management of pediatric low grade gliomas. Int J Radiat Oncol Biol Phys. 2001 Nov 1;51(3):704-10. doi: 10.1016/s0360-3016(01)01705-9. PMID 11597812
- [Background] Duffner PK, Horowitz ME, Krischer JP, Friedman HS, Burger PC, Cohen ME, Sanford RA, Mulhern RK, James HE, Freeman CR, et al. Postoperative chemotherapy and delayed radiation in children less than three years of age with malignant brain tumors. N Engl J Med. 1993 Jun 17;328(24):1725-31. doi: 10.1056/NEJM199306173282401. PMID 8388548
- [Background] Brown MT, Friedman HS, Oakes WJ, Boyko OB, Hockenberger B, Schold SC Jr. Chemotherapy for pilocytic astrocytomas. Cancer. 1993 May 15;71(10):3165-72. doi: 10.1002/1097-0142(19930515)71:103.0.co;2-n. PMID 8490847
- [Background] Gajjar A, Bhargava R, Jenkins JJ, Heideman R, Sanford RA, Langston JW, Walter AW, Kuttesch JF, Muhlbauer M, Kun LE. Low-grade astrocytoma with neuraxis dissemination at diagnosis. J Neurosurg. 1995 Jul;83(1):67-71. doi: 10.3171/jns.1995.83.1.0067. PMID 7782852
- [Background] Ceppa EP, Bouffet E, Griebel R, Robinson C, Tihan T. The pilomyxoid astrocytoma and its relationship to pilocytic astrocytoma: report of a case and a critical review of the entity. J Neurooncol. 2007 Jan;81(2):191-6. doi: 10.1007/s11060-006-9216-z. Epub 2006 Jul 19. PMID 16850101
- [Background] Tsugu H, Oshiro S, Yanai F, Komatsu F, Abe H, Fukushima T, Nomura Y, Matsumoto S, Nabeshima K, Takano K, Utsunomiya H. Management of pilomyxoid astrocytomas: our experience. Anticancer Res. 2009 Mar;29(3):919-26. PMID 19414328
- [Background] Lefkowitz IB, Packer RJ, Sutton LN, Siegel KR, Bruce DA, Evans AE, Schut L. Results of the treatment of children with recurrent gliomas with lomustine and vincristine. Cancer. 1988 Mar 1;61(5):896-902. doi: 10.1002/1097-0142(19880301)61:53.0.co;2-c. PMID 3338054
- [Background] Petronio J, Edwards MS, Prados M, Freyberger S, Rabbitt J, Silver P, Levin VA. Management of chiasmal and hypothalamic gliomas of infancy and childhood with chemotherapy. J Neurosurg. 1991 May;74(5):701-8. doi: 10.3171/jns.1991.74.5.0701. PMID 1901597
- [Background] Friedman HS, Krischer JP, Burger P, Oakes WJ, Hockenberger B, Weiner MD, Falletta JM, Norris D, Ragab AH, Mahoney DH Jr, et al. Treatment of children with progressive or recurrent brain tumors with carboplatin or iproplatin: a Pediatric Oncology Group randomized phase II study. J Clin Oncol. 1992 Feb;10(2):249-56. doi: 10.1200/JCO.1992.10.2.249. PMID 1732426
- [Background] Packer RJ, Sutton LN, Bilaniuk LT, Radcliffe J, Rosenstock JG, Siegel KR, Bunin GR, Savino PJ, Bruce DA, Schut L. Treatment of chiasmatic/hypothalamic gliomas of childhood with chemotherapy: an update. Ann Neurol. 1988 Jan;23(1):79-85. doi: 10.1002/ana.410230113. PMID 3345069
- [Background] Janss AJ, Grundy R, Cnaan A, Savino PJ, Packer RJ, Zackai EH, Goldwein JW, Sutton LN, Radcliffe J, Molloy PT, et al. Optic pathway and hypothalamic/chiasmatic gliomas in children younger than age 5 years with a 6-year follow-up. Cancer. 1995 Feb 15;75(4):1051-9. doi: 10.1002/1097-0142(19950215)75:43.0.co;2-s. PMID 7842408
- [Background] Sievert AJ, Fisher MJ. Pediatric low-grade gliomas. J Child Neurol. 2009 Nov;24(11):1397-408. doi: 10.1177/0883073809342005. PMID 19841428
- [Background] Burkhard C, Di Patre PL, Schuler D, Schuler G, Yasargil MG, Yonekawa Y, Lutolf UM, Kleihues P, Ohgaki H. A population-based study of the incidence and survival rates in patients with pilocytic astrocytoma. J Neurosurg. 2003 Jun;98(6):1170-4. doi: 10.3171/jns.2003.98.6.1170. PMID 12816259
- [Background] Wallner KE, Gonzales MF, Edwards MS, Wara WM, Sheline GE. Treatment results of juvenile pilocytic astrocytoma. J Neurosurg. 1988 Aug;69(2):171-6. doi: 10.3171/jns.1988.69.2.0171. PMID 3392563
- [Background] Mamelak AN, Prados MD, Obana WG, Cogen PH, Edwards MS. Treatment options and prognosis for multicentric juvenile pilocytic astrocytoma. J Neurosurg. 1994 Jul;81(1):24-30. doi: 10.3171/jns.1994.81.1.0024. PMID 8207524
- [Background] Dutton JJ. Gliomas of the anterior visual pathway. Surv Ophthalmol. 1994 Mar-Apr;38(5):427-52. doi: 10.1016/0039-6257(94)90173-2. PMID 8009427
- [Background] Opocher E, Kremer LC, Da Dalt L, van de Wetering MD, Viscardi E, Caron HN, Perilongo G. Prognostic factors for progression of childhood optic pathway glioma: a systematic review. Eur J Cancer. 2006 Aug;42(12):1807-16. doi: 10.1016/j.ejca.2006.02.022. Epub 2006 Jun 30. PMID 16809032
- [Background] Cappelli C, Grill J, Raquin M, Pierre-Kahn A, Lellouch-Tubiana A, Terrier-Lacombe MJ, Habrand JL, Couanet D, Brauner R, Rodriguez D, Hartmann O, Kalifa C. Long-term follow up of 69 patients treated for optic pathway tumours before the chemotherapy era. Arch Dis Child. 1998 Oct;79(4):334-8. doi: 10.1136/adc.79.4.334. PMID 9875044
- [Background] Silva MM, Goldman S, Keating G, Marymont MA, Kalapurakal J, Tomita T. Optic pathway hypothalamic gliomas in children under three years of age: the role of chemotherapy. Pediatr Neurosurg. 2000 Sep;33(3):151-8. doi: 10.1159/000028996. PMID 11096362
- [Background] Nicholson HS, Kretschmar CS, Krailo M, Bernstein M, Kadota R, Fort D, Friedman H, Harris MB, Tedeschi-Blok N, Mazewski C, Sato J, Reaman GH. Phase 2 study of temozolomide in children and adolescents with recurrent central nervous system tumors: a report from the Children's Oncology Group. Cancer. 2007 Oct 1;110(7):1542-50. doi: 10.1002/cncr.22961. PMID 17705175
- [Background] Gil-Grande LA, Boixeda D, Garcia-Hoz F, Barcena R, Lledo A, Suarez E, Pascasio JM, Moreira V. Treatment of liver hydatid disease with mebendazole: a prospective study of thirteen cases. Am J Gastroenterol. 1983 Sep;78(9):584-8. PMID 6613972
- [Background] Bai RY, Staedtke V, Aprhys CM, Gallia GL, Riggins GJ. Antiparasitic mebendazole shows survival benefit in 2 preclinical models of glioblastoma multiforme. Neuro Oncol. 2011 Sep;13(9):974-82. doi: 10.1093/neuonc/nor077. Epub 2011 Jul 15. PMID 21764822
- [Background] Mukhopadhyay T, Sasaki J, Ramesh R, Roth JA. Mebendazole elicits a potent antitumor effect on human cancer cell lines both in vitro and in vivo. Clin Cancer Res. 2002 Sep;8(9):2963-9. PMID 12231542
- [Background] Sasaki J, Ramesh R, Chada S, Gomyo Y, Roth JA, Mukhopadhyay T. The anthelmintic drug mebendazole induces mitotic arrest and apoptosis by depolymerizing tubulin in non-small cell lung cancer cells. Mol Cancer Ther. 2002 Nov;1(13):1201-9. PMID 12479701
- [Background] Doudican N, Rodriguez A, Osman I, Orlow SJ. Mebendazole induces apoptosis via Bcl-2 inactivation in chemoresistant melanoma cells. Mol Cancer Res. 2008 Aug;6(8):1308-15. doi: 10.1158/1541-7786.MCR-07-2159. Epub 2008 Jul 30. PMID 18667591
- [Background] Dobrosotskaya IY, Hammer GD, Schteingart DE, Maturen KE, Worden FP. Mebendazole monotherapy and long-term disease control in metastatic adrenocortical carcinoma. Endocr Pract. 2011 May-Jun;17(3):e59-62. doi: 10.4158/EP10390.CR. PMID 21454232
- [Background] Vutova K, Mechkov G, Vachkov P, Petkov R, Georgiev P, Handjiev S, Ivanov A, Todorov T. Effect of mebendazole on human cystic echinococcosis: the role of dosage and treatment duration. Ann Trop Med Parasitol. 1999 Jun;93(4):357-65. doi: 10.1080/00034989958357. PMID 10656037
- [Background] Kepes JJ, Rubinstein LJ, Eng LF. Pleomorphic xanthoastrocytoma: a distinctive meningocerebral glioma of young subjects with relatively favorable prognosis. A study of 12 cases. Cancer. 1979 Nov;44(5):1839-52. doi: 10.1002/1097-0142(197911)44:53.0.co;2-0. PMID 498051
- [Background] Rao AA, Laack NN, Giannini C, Wetmore C. Pleomorphic xanthoastrocytoma in children and adolescents. Pediatr Blood Cancer. 2010 Aug;55(2):290-4. doi: 10.1002/pbc.22490. PMID 20582976
- [Background] Giannini C, Scheithauer BW, Burger PC, Brat DJ, Wollan PC, Lach B, O'Neill BP. Pleomorphic xanthoastrocytoma: what do we really know about it? Cancer. 1999 May 1;85(9):2033-45. PMID 10223246